CLINICAL TRIAL: NCT01303770
Title: Development and Evaluation of a Cognitive Rehabilitation Program for Persons With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Eynat Shevil, Dr. Eynat Shevil, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MSCogRehab; PIRG03-GA-2008-230959 (Other Grant/Funding Number: European Commission FP7 Marie Curie IRG)
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Multiple Sclerosis; Cognitive Impairment
Keywords: Multiple Sclerosis; Cognitive impairment; Self-management programs; Occupational Therapy; Rehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Cognitive intervention group (Experimental): Cognitive rehabilitation program designed to be tested in this study
  Interventions: Behavioral: Self-management cognitive rehabilitation group intervention
- Control group (Active Comparator)
  Interventions: Behavioral: Control intervention

INTERVENTIONS:
Behavioral: Self-management cognitive rehabilitation group intervention — 8-week cognitive rehabilitation program facilitated by an occupational therapist. Program goals include increased knowledge of cognitive impairments in multiple sclerosis, increased self-efficacy to manage cognitive changes and increased use of cognitive compensatory strategies.
  Arms: Cognitive intervention group
Behavioral: Control intervention — 8-week group program that is not specifically directed to management of cognitive impairments.
  Arms: Control group

SUMMARY:
Multiple sclerosis (MS) is a progressive neurological disease that affects over 2.5 million people worldwide. Up to 50% of persons with MS (PwMS) will experience some form of cognitive impairment as a result of the disease including disturbances in memory, attention, concentration, information processing, and executive functions such as problem solving, and self-monitoring. MS-related cognitive impairments negatively affect many aspects of functioning and independent participation in everyday life. Thus, PwMS who experience cognitive impairments face a wide array of recurring barriers that pose grave challenges to carrying out everyday activities while trying to maintain multiple life roles and as they age.

Management of cognitive symptoms can be addressed through rehabilitation which has the potential to reduce disability, prevent complications of the disease, and enhance participation, independence, and quality of life. Considering the high frequency of cognitive impairments in MS and their significant, complex impact on functioning and independence, it is critical that cognitive interventions be an essential component of MS rehabilitation.

The overarching goal of this study is to develop and test a self-management, group-based cognitive rehabilitation program designed specifically for PwMS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS
* 18 years of age or older
* Self-report of cognitive difficulties

Exclusion Criteria:

* Exacerbation of symptoms in past 3 months
* History of TBI, CVA, epilepsy, Psychiatric condition, drug/alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive strategy use | pre intervention, post intervention, 3,6,12 month followup

SECONDARY OUTCOMES:
Cognitive self-efficacy | pre-intervention, post intervention, 3,6,12 month followup

CONTACTS AND LOCATIONS:
Overall Officials: Eynat Shevil, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Rabin Medical Center, Multiple Sclerosis Clinic, Petah Tikva, Israel